CLINICAL TRIAL: NCT02080208
Title: Which Place for High Flow Oxygen in Intensive Care Unit ?
Brief Title: Which Place for High Flow Oxygen in ICU ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Bialais, physiotherapist PhD student, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: OptSCM
Record Dates: First submitted 2014-01-09; First posted 2014-03-06 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Hypoxemia
Keywords: hypoxemia; high flow oxygen therapy; respiratory failure
MeSH Terms: conditions — Hypoxia; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flow Oxygen (Experimental): Patients receiving oxygen via high flow oxygen therapy (Optiflow)
  Interventions: Device: Optiflow
- Conventionnal (No Intervention): patients receiving oxygen via conventional way (low flow)

INTERVENTIONS:
Device: Optiflow — patients receive oxygen via high flow oxygen therapy during 20 minutes
  Arms: High Flow Oxygen

SUMMARY:
Patients with respiratory failure often need oxygen and/or ventilatory support. Patients who need only oxygen support, usually received low flow oxygen (< 15 Liters / min), as well as in respiratory weaning. Now new devices can be used. They provide high flow oxygen with different benefits. This high flow devices provide exact fraction of inspired oxygen (FiO2), allows a positive end expiratory pressure and supplies a wash out flow. The hypothesis of this study is that the high flow oxygen enable more efficient oxygen administration than conventional oxygen. In addition, it would improve the effectiveness of the ventilation of the patient, through flushing the dead space.

DETAILED DESCRIPTION:
The investigators hypothesized that when using high flow oxygen therapy, respiratory failure is relieved, as well as ventilation failure, so accessories are less stressed muscles, and this can be demonstrated by the electromyography (EMG) of sterno-mastoid..

ELIGIBILITY:
Inclusion Criteria: patients with respiratory failure.

* Spontaneously breathing patient requiring administration at least 40% oxygen, or,
* Patient under mechanical ventilation, during respiratory weaning.

Exclusion Criteria:

* Facial trauma, active hemoptysis, pneumothorax, thoraco-abdominal surgery or upcoming intubation for spontaneously breathing patients.
* Neuromuscular disease, altered consciousness or agitation for patients under mechanical ventilation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Oxygenation criteria | 20 minutes
  Arterial oxygen partial pressure (PO2), oxygen saturation by pulse oximetry (SpO2), arterial PO2/FiO2, positive end expiratory pressure (PEEP)

SECONDARY OUTCOMES:
Change from baseline in Ventilation criteria | 20 minutes
  respiratory rate (RR), arterial partial CO2 pressure (PCO2), pH, sterno-mastoid EMG

OTHER OUTCOMES:
change from baseline in hemodynamic criteria | 20 minutes
  cardiac frequency, arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Bialais, PhD Student, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No